CLINICAL TRIAL: NCT02635074
Title: A Phase I Dose Escalation Study of Ibrutinib With Idarubicin/Cytarabine for Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Ibrutinib, Idarubicin and Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: safety
Sponsor: Steven E. Coutre (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Steven E. Coutre, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEMAML0036; NCI-2015-01961 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 35003; IRB-35003 (Other: Stanford IRB); P30CA124435 (NIH)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; ibrutinib; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, idarubicin, cytarabine) (Experimental): INDUCTION: Ibrutinib daily on days 1 to 21, idarubicin intravenously (IV) over 15 minutes on days 1 to 3 and cytarabine IV continuously on days 1 to 4.
  CONSOLIDATION: Patients achieving CR or CRi may receive ibrutinib daily on days 1 to 21, idarubicin IV over 15 minutes on days 1 to 2 and cytarabine IV continuously on days 1 to 3. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients maintaining a CR/CRi may receive ibrutinib daily on days 1 to 28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Ibrutinib; Drug: Idarubicin

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: Beta-cytosine arabinoside; 1-beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-beta-D-arabinofuranosylcytosine; 2(1H)-pyrimidinone, 4-amino-1-beta-d-arabinofuranosyl; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Ibrutinib — Given PO
  Other Names: Imbruvica; BTK Inhibitor PCI-32765; PCI-32765; CRA-032765
Drug: Idarubicin — Given IV
  Other Names: Idamycin; Zavedos; 4-Demethoxydaunomycin; 4-Demethoxydaunorubicin; 4-DMDR

SUMMARY:
This phase I trial studies the side effects and best dose of ibrutinib when given together with idarubicin and cytarabine in treating patients with acute myeloid leukemia that has returned after a period of improvement or has not responded to previous treatment. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ibrutinib together with idarubicin and cytarabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Identify the safety and recommended phase 2 dose of ibrutinib in combination with idarubicin/cytarabine in relapsed/refractory acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

* Assess the induction response rate (complete remission [CR]/complete remission with incomplete count [CRi]) of ibrutinib in combination with idarubicin/cytarabine in relapsed/refractory AML.
* Assess overall survival of ibrutinib in combination with idarubicin/cytarabine in relapsed/refractory AML.

OUTLINE: This is a dose-escalation study of ibrutinib.

INDUCTION: Patients receive ibrutinib orally (PO) once daily (QD) on days 1 to 21, idarubicin intravenously (IV) over 15 minutes on days 1 to 3 and cytarabine IV continuously on days 1 to 4.

CONSOLIDATION: Patients achieving CR or CRi may receive ibrutinib PO QD on days 1 to 21, idarubicin IV over 15 minutes on Days 1and 2 and cytarabine IV continuously on days 1-3. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients maintaining a CR/CRi may receive ibrutinib PO QD on days 1 to 28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
INCLUSION CRITERIA

* Previous morphologically-confirmed diagnosis of acute myeloid leukemia (AML) based on World Health Organization (WHO) Criteria
* At least one prior chemotherapy regimen to treat AML
* Disease relapse or refractory disease as shown by > 5% blasts in the bone marrow (not attributable to another cause). Administration of hydrea to control high WBC count is permitted.
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, or Karnofsky Performance Status (KPS) ≥ 60%
* Life expectancy > 4 weeks
* Platelet count ≥ 10,000/mm3 within 72 hours of initiating the Induction Cycle (platelet transfusion support is allowed)
* Serum creatinine ≤ 2.0 mg/dL within 72 hours of initiating the Induction Cycle
* Total bilirubin ≤ 2.1 mg/dL within within 72 hours of initiating the Induction Cycle (EXCEPTION: If elevation is not due to liver dysfunction, and is due primarily to elevated unconjugated hyperbilirubinemia secondary to Gilbert's syndrome, or hemolysis of non-hepatic origin)
* Serum glutamic oxaloacetic transaminase (SGOT) [aspartate aminotransferase (AST) ] ≤ 3.0 X upper limit of normal (ULN) within 72 hours of initiating the Induction Cycle
* Serum glutamic pyruvic transaminase (SGPT) [alanine aminotransferase (ALT)] ≤ 3.0 X ULN within 72 hours of initiating the Induction Cycle
* Baseline prothrombin time (PT)/international normalized ratio (INR) ratio < 3 X ULN within 7 days of initiating the Induction Cycle (for subjects with correctable coagulation abnormalities, coagulation factor support per institutional standard of care for AML is allowed)
* Partial thromboplastin time (PTT) < 3 X ULN within 7 days of initiating the Induction Cycle (for subjects with correctable coagulation abnormalities, coagulation factor support per institutional standard of care for AML is allowed)
* Negative pregnancy test within 14 days prior to study treatment (for Women of reproductive potential only)
* Women of child-bearing potential and men must agree (in ICF) to use adequate contraception (eg, hormonal or barrier methods of birth control; abstinence; sterilized partner) for the duration of study participation
* Ability to understand and the willingness to sign the written informed consent document

EXCLUSION CRITERIA

* Received anticancer therapy (chemotherapy, immunotherapy, radiotherapy, or investigational therapy) within 2 weeks prior to starting study treatment [EXCEPTION: Hydroxyurea (hydrea) to control high white blood cell count is permitted]
* Receiving any other investigational agents within 14 days or 5 effective half lives (whichever is shorter) prior to 1st dose of ibrutinib
* Prior treatment with ibrutinib
* Known unresolved toxicities due to prior anticancer therapy [≥ Grade 2, by Common Terminology Criteria for Adverse Events (CTCAE) v4.03] unless otherwise defined in the inclusion/exclusion criteria (EXCEPTION: alopecia)
* Known acute promyelocytic leukemia (French-American-British Class M3-AML)
* Known active central nervous system (CNS) leukemia
* Prior bone marrow transplant presenting with active uncontrolled graft vs host disease (GvHD)
* Known congenital bleeding disorders, such as hemophilia
* Known history of stroke or intracranial hemorrhage within 6 months prior to study treatment
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with strong CYP3A inhibitors at the time of study enrollment. Washout period is 5 effective half-lives is required prior to 1st dose of ibrutinib
* Requires treatment with strong CYP3A inducers at the time of study enrollment. Washout period is 5 effective half-lives is required prior to 1st dose of ibrutinib
* Known active uncontrolled systemic infection
* Major surgery within 4 weeks of 1st dose of ibrutinib
* Unable to swallow capsules
* Known Malabsorption syndrome
* Known Disease significantly affecting gastrointestinal function
* Resection of the stomach or small bowel
* Uncontrolled symptomatic inflammatory bowel disease
* Ulcerative colitis
* Bowel obstruction, partial or complete
* Congestive heart failure with ejection fraction (EF) < 45%
* Uncontrolled cardiac disease, including uncontrolled cardiac arrhythmia or coronary artery disease (CAD) with active symptoms due to CAD defined as unstable angina
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib; idarubicin; or cytarabine
* Uncontrolled intercurrent illness including, but not limited to:
* Active infection
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant
* Lactating
* Known positive HIV
* Known active hepatitis C
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07-18 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Induction Response Rate | 12 weeks
  The induction Response Rate (CR/CRi) of ibrutinib in combination with idarubicin/cytarabine in relapsed/refractory AML was assessed as the number of participants who achieving a complete response (CR) or complete response with incomplete blood count recovery (CRi), divided by the total number of participants completing induction therapy.

SECONDARY OUTCOMES:
Overall Survival (OS) | 6 months
  Overall survival (OS) was assessed as the number of patients remaining alive 6 months after the initiation of study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Steven Coutre, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States